CLINICAL TRIAL: NCT03403920
Title: Validity of the Turkish Version of the Profile Fitness Mapping Low Back Questionnaire for Patients With Low Back Pain
Brief Title: Validity of Profile Fitness Mapping Low Back Questionnaire
Status: Completed | Type: Observational
Sponsor: HATİCE ÇETİN (Other)
Responsible Party: Sponsor-Investigator, HATİCE ÇETİN, Research Assistant, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: 7763482
Record Dates: First submitted 2018-01-08; First posted 2018-01-19 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain; Pain; Assessment, Self; Disability Physical
Keywords: validity; low back pain; functional; pain; questionnaire
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Profile Fitness Mapping Low Back Questionnaire

SUMMARY:
As patients improve on one parametric result, the results on the other parametric may worsen, but the total score may not be affected. For this reason, it would be useful to make measurements that evaluate all the parameters of the patients. Thus, it would be more advantageous to score both pain and symptoms separately, as well as activity limitations. Therefore, neck specific surveys are needed to meet this need.

For this reason, this study was planned to determine the validity of the questionnaire named "Profile Fitness Mapping Low Back Questionnaire" in patients with low back pain.

DETAILED DESCRIPTION:
The translation of the original version of "Profile Fitness Mapping Low Back Questionnaire" to Turkish will be translated by two independent professional translators. Afterwards, a person without a medical history and a native English speaker will be translated into English again. Once the translation stages are complete, the translators will be brought together to discuss the two versions of the questionnaire. Then the final state will be translated into the main language of the questionnaire and the compliance will be checked.

First of all, people who have been suffering from low back pain for at least six months will complete the "Profile Fitness Mapping Low Back Questionnaire", "Oswestry Disability Index" and "SF-36 health related quality of life questionnaire".

Seven days after the questionnaire, the "Profile Fitness Mapping Low Back Questionnaire" will be completed again.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for more than six months during activity or rest
* Having a problem with low back based on clinical examination and story

Exclusion Criteria:

* Having neurological problems
* Having vestibular or cerebellar problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have neck pain more than six months
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Profile Fitness Mapping Low Back Questionnaire | Change from Baseline Profile Fitness Mapping Low Back Questionnaire score (functional limitation and symptom score) at 1 week.
  The Profile Fitness Mapping Low Back Questionnaire was developed between 1992 and 1994 at the Alfta Rehab Center and consists of two back specific scales, designed for the assessment of self-estimated symptoms and functional limitations. The symptom scale contains two indices of separate aspects of symptomatology. All items are given six response alternatives (how often: range from 1 = never/very seldom, to 6 = very often/always; how much: range from 7 = nothing/none at all, to 12 = almost unbearable/ unbearable, all/maximally).The functional limitation scale (one index) and the symptom scale (two indices) are presented in a self-administered form. All items were given six response alternatives (ranging from
  1 = very good, no problem, very satisfying, very likely, to 6 = very bad, very difficult/impossible, very dissatisfying, very unlikely). Higher index scores reflect better function/better health.

SECONDARY OUTCOMES:
Oswestry Disability Index | All of the participants will assess at baseline with this index.
  The Oswestry Disability Index assesses ten different aspects of disability (pain, personal care, lifting, sitting, standing, sleeping, sex life, social life, walking and travelling). Each parameter is scored from 0 to 5, with 0 indicating no functional limitation due to pain and 5 indicating a major functional disability due to low back pain. This questionnaire is scored using a global percentage score. The obtainable maximum score is 50, which corresponds to 100%. A score of 0%-20% means minimal disability, 21%-40% means moderate disability, 41%-60% means severe disability, 61%-80% means crippling back pain, and 81%-100% means bed-bound or exaggerated symptoms.
SF-36 health related quality of life questionnaire | All of the participants will assess at baseline with this questionnaire.
  The SF-36 questionnaire consists of 36 items, which are used to calculate eight subscales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The first four scores can be summed to create the physical composite score, while the last four can be summed to create the mental composite score. Scores for the SF-36 scales range between 0 and 100, with higher scores indicating a better quality of life.
Visual Analog Scale | All of the participants will assess at baseline with this scale.
  The pain Visual Analog Scale is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorklund M, Hamberg J, Heiden M, Barnekow-Bergkvist M. The assessment of symptoms and functional limitations in low back pain patients: validity and reliability of a new questionnaire. Eur Spine J. 2007 Nov;16(11):1799-811. doi: 10.1007/s00586-007-0405-z. Epub 2007 Jun 22. PMID 17587068